CLINICAL TRIAL: NCT01980186
Title: Transcranial Ultrasonography Using Linear 2D Imaging of the Brain and Surrounding Tissues
Brief Title: Transcranial Ultrasonography Using Linear 2D Imaging of the Brain
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Brain Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: BTC-002
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Autism; Extra-axial Fluid
Keywords: transcranial ultrasound; autism; cortical dysplasia; extra-axial fluid
MeSH Terms: conditions — Autistic Disorder; Malformations of Cortical Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Individuals with autism: Both individuals with autism and their siblings will be evaluated with (TUS)transcranial 2D ultrasound.
  Interventions: Device: TUS transcranial 2D ultrasound
- Siblings of individuals with autism: Non-autistic siblings with no other obvious health issues will be screened
  Interventions: Device: TUS transcranial 2D ultrasound

INTERVENTIONS:
Device: TUS transcranial 2D ultrasound

SUMMARY:
This study will use linear 2D ultrasound imaging to look at the brain of individuals diagnosed with autism and their siblings. This is called transcranial ultrasound (TUS). It is hypothesized that TUS will allow real-time imaging of the fluid spaces outside the brain and will further allow the imagining of brain areas important to language and social function.

DETAILED DESCRIPTION:
TUS will be evaluated as a simple and low cost screening technique to evaluate the presence of increased extra-axial fluid (EAF)or(subarachnoid cerebral spinal fluid). A recent study (Shen et al. 2013) demonstrated increased EAF was predictive of risk of autism. We believe TUS is capable or rapid, safe, low cost, non-invasive measurement of EAF spaces. Where prior imaging, ie., MRI or CT exist they will be used as comparisons. Both individuals with autism and their siblings will be screened to create a database and standard for TUS measurements. It is further believed that TUS may be able to detect areas of cortical abnormalities called dysplasias. The procedure requires no sedation and only takes a few minutes to perform. If validated, this would make TUS an ideal screening test for autism risk and allow for early referral and more definitive imaging with MRI where necessary.

ELIGIBILITY:
Inclusion Criteria: Confirmed diagnosis of autism or the sibling thereof and willingness of a parent to consent and where applicable for the individual to assent or consent depending on age.

-

Exclusion Criteria: Siblings must have no obvious health issues or developmental abnormalities.

-

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with autism of any age and their neurotypical otherwise healthy siblings of any included age (6 months to 21 years).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Extra-axial fluid as measured at the gyral summit. | This study will collect data for up to 3 years to determine the accuracy of the predictive assessments for autism risk
  TUS is performed with linear 2D acoustical outputs in the 10-5MHz range. These are typical for TUS investigations with doppler and the only difference is the linear output of the probe.

CONTACTS AND LOCATIONS:
Overall Officials: James J Bradstreet, MD, Principal Investigator — Brain Treatment Center
Locations (2):
- United States (2):
  - Brain Treatment Center, Newport Beach, California
  - Brain Treatment Center, Buford, Georgia